CLINICAL TRIAL: NCT00424645
Title: Randomized, Double-Blind, Placebo Controlled Trial of Voraxaze™ in Patients With a Delayed MTX Clearance
Brief Title: Voraxaze for Delayed Methotrexate Clearance
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated due to low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2006-0119
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hematologic Malignancy; Solid Tumor
Keywords: Hematologic Malignancy; Solid Tumor; Glucarpidase; Voraxaze; Delayed Methotrexate Clearance; Placebo
MeSH Terms: conditions — Hematologic Neoplasms | interventions — glucarpidase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voraxaze (Experimental): Voraxaze administered 50 units/kg intravenously (IV) repeated a maximum of 2 times in a given cycle of chemotherapy.
  Interventions: Drug: Voraxaze (Glucarpidase)
- Placebo (Placebo Comparator): Placebo administered IV following Voraxaze arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voraxaze (Glucarpidase) — 50 units/kg IV within 12 hours of study eligibility being confirmed.
  Other Names: Carboxypeptidease
  Arms: Voraxaze
Drug: Placebo — Administered by IV within 12 hours of study eligibility being confirmed.
  Arms: Placebo

SUMMARY:
Primary Objectives:

1. To evaluate the efficacy of Glucarpidase (Voraxaze) in increasing the rate of methotrexate (MTX) clearance following high dose MTX treatment in patients with a delayed MTX clearance.
2. To evaluate the pharmacokinetics (PK) of Glucarpidase following high dose MTX treatment in patients with a delayed MTX clearance.
3. To evaluate the safety profile of Glucarpidase following high dose MTX treatment in patients with a delayed MTX clearance.

Secondary Objectives:

1. To evaluate the effect of Glucarpidase on the incidence of neutropenic fever and use of intravenous (IV) antibiotics.
2. To evaluate the effect of Glucarpidase on the length of hospitalization.
3. To evaluate the effect of Glucarpidase on renal function.
4. To evaluate the effect of Glucarpidase on Quality of Life (QOL).
5. To evaluate the anti-glucarpidase antibody response.
6. To evaluate the efficacy of Glucarpidase following its use in repeated cycles of high dose MTX treatment.

DETAILED DESCRIPTION:
Researchers want to learn how glucarpidase may impact patients' length of stay in the hospital, kidney function, and quality of life. Also, researchers want to learn if glucarpidase may decrease the incidence of neutropenic fever, which may decrease the use of antibiotics by vein to treat this kind of fever.

MTX is a high-dose chemotherapy drug that reduces the supply of an important vitamin (folate) required for the growth of cancer cells. In patients with delayed clearance of MTX from the body, there is a risk of more frequent or severe side effects from the drug.

Glucarpidase is a drug that breaks down MTX in the blood, causing the drug to be less toxic and decreasing levels of the drug in the blood.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded. You will have a physical exam, including measurement of your vital signs (temperature, pulse, breathing rate, and blood pressure). You will have blood drawn (about 3 teaspoons) for routine tests. You will also have blood drawn (about 1 teaspoon), right before treatment starts, 28 days after the first dose of study drug in each cycle, and at the end of the study to see if you have any antibodies (proteins in the body that help fight infections and foreign substances in the body) to the study drug. Women who are able to have children must have a negative blood pregnancy test. The blood used for the pregnancy test will come from the sample taken for routine tests. (There is no additional blood draw for the pregnancy test).

You may be given either glucarpidase or placebo (a drug that looks like glucarpidase but is not active). Neither you nor the study doctor will know if you have been given glucarpidase or placebo. This is called the blinded phase of this study. Before you can begin on this study, if you are already suffering from side effects (because of difficulty with MTX clearance), such as kidney toxicity, severe mucositis (redness and painful ulcers in the mouth), and/or you have extremely high MTX levels, you will not be randomized and will receive glucarpidase, not placebo. If this is the case, your doctor will know that you have been given glucarpidase.

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 treatment groups, which will be based on the dose of MTX you received. You will then be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive glucarpidase. Participants in the other group will receive placebo. There is a higher chance that you may receive glucarpidase than placebo because for every patient that receives placebo, 2 patients will receive glucarpidase. The glucarpidase or placebo dose that you may receive will be given by vein within 12 hours after you have been found eligible to participate in this study. Glucarpidase or placebo will be given during the first study cycle (after MTX treatment is completed, if after 72 hours your MTX levels are found to be high). You may receive additional doses of glucarpidase (depending upon the level of MTX in your blood) up to a maximum of 2 doses. If this is the case, the second dose will be given at least 24 hours after the first dose you received.

Regardless of the treatment group that you are assigned to, you will continue to receive standard treatment (fluids by vein with sodium acetate or sodium bicarbonate and leucovorin) for high MTX levels. In future cycles of MTX, you may receive glucarpidase, if you continue to experience a delay of MTX clearing from your body. The glucarpidase dose may be repeated a maximum of 2 times in a given cycle of chemotherapy. The length of a cycle of chemotherapy will vary, depending on the dose of MTX and the regimen the patient is receiving. One cycle of treatment with glucarpidase is at least 24 hours apart.

You will be asked to fill out several questionnaires regarding your quality of life. These questionnaires will ask about your level of pain, fatigue, nausea, sleep disturbances, etc. They will be given during the first study cycle only (before the study drug is given and daily during the first study cycle). They will take about 5 minutes to complete each time.

You will also have blood drawn (about 3 teaspoons each), at different times, so that study doctors can monitor your kidney function and liver function, depending on your clinical condition. These blood samples will be drawn at least twice a week while you are on this study. You will again have blood drawn for the presence of antibodies 14 days after treatment with glucarpidase, before every cycle of MTX treatment, and at the end of this study.

You will be taken off this study if your disease gets worse, you experience intolerable side effects, or you completed planned therapy (a maximum of 6 cycles of study drug). At the end of this study, your complete medical history will again be recorded. You will have a physical exam, including measurement of your vital signs. You will also have blood drawn (about 1 teaspoon) for routine tests.

This is an investigational study. Glucarpidase is not FDA approved or commercially available. The M. D. Anderson Institutional Review Board (IRB) has authorized the use of glucarpidase for research only. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. Glucarpidase and placebo will be provided free of charge during this study. Up to 46 patients will take part in this study. All patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with solid tumors and hematologic malignancies, receiving high dose methotrexate (MTX) (> / = 1 g/m^2 up to 14 g/m^2), who have delayed MTX clearance. Delayed MTX clearance is defined as: a) Serum MTX level at 72 +/- 2 hrs from initiation of infusion > / = 0.1 µmol/L for MTX doses 1-3.5 g/m^2 OR b) Serum MTX level at 72 +/- 2 hrs from initiation of infusion > / = 0.3 µmol/L for MTX doses > 3.5 g/m^2
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. IRB-approved signed informed consent

Exclusion Criteria:

1. Any medical or psychiatric illness that is deemed by the investigator to be likely to interfere with patient's ability to sign informed consent, cooperate and participate in the study
2. Patients receiving medications which may interfere with MTX excretion or enhance MTX toxicity (e.g. Penicillins, Cephalosporins, Tetracyclines, Non-Steroidal Anti-inflammatory Agents, Salicylates, Thiazide Diuretics, Bactrim, and Probenecid)
3. Patients with uncontrolled cardiac disease such as uncontrolled angina, cardiac arrhythmia, or Congestive Heart Failure (CHF) (New York Heart Association (NYHA) 4)
4. Patients with known hypersensitivity to any of the components of the study drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 01/09/07 through 01/31/08. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study closed early by sponsor due to low accrual. Of three patients enrolled, only two patients received blinded study drug. Study terminated prior to other randomization.
Period: Overall Study
Arm/Group | Voraxaze | Placebo
Started | 3 | 0
Completed | 2 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voraxaze | Placebo | Total
Number analyzed (Participants) | 3 | 0 | 3
Age Continuous [Mean (Full Range); unit: years] | 64 [46 to 72] |  | 64 [46 to 72]
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 3 |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Response Rate (Percentage)
Description: Response rate defined as proportion of patients that clear methotrexate (MTX) at 15 min and 24-hour post infusion of study drug, Glucarpidase (Voraxaze) to total patient number. Serum MTX levels (standard methods and mass spectrometry) at 15 minutes, 24 hours, or daily until MTX clearance defined as serum MTX level <0.1 µmol/L.
Time Frame: Study period 2 years
Population: Analysis was to be per protocol, low accrual and early termination led too few responses for evaluation.
Arm/Group | Voraxaze | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Voraxaze | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voraxaze (N=3) | Placebo (N=0)
Fever with Hypotension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No